CLINICAL TRIAL: NCT00374920
Title: A Multicenter, Double Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of MEM 1003 for the Treatment of Patients With Bipolar I Disorder Suffering Acute Manic or Mixed Episodes
Brief Title: Safety and Efficacy of MEM 1003 Versus Placebo for the Treatment of Patients With Bipolar I Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memory Pharmaceuticals (Industry)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Amy S. Domanowski, Ph.D., Head Regulatory Affairs, Memory Pharmaceuticals Corp.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEM 1003-101
Record Dates: First submitted 2006-09-09; First posted 2006-09-12 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Bipolar Disorder With Manic or Mixed Episodes
Keywords: bipolar; mania; mixed
MeSH Terms: conditions — Mania

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MEM 1003

SUMMARY:
The purpose of this study is to establish the potential of MEM 1003 as a safe and effective treatment for patients with an acute manic or mixed episode of bipolar disorder.

DETAILED DESCRIPTION:
Bipolar affective disorder is one of the most common, severe, and persistent mental illnesses. It is characterized by periods of deep, prolonged, and profound depressions that alternate with periods of excessively elevated and/or irritable mood (mania). The pathophysiology of bipolar disorder is complex, and can include an inheritable component, administration of antidepressant medications, behavioral sensitization processes, and neuronal calcium dysregulation that leads to apoptosis of critical brain circuitry that regulates emotion. Addressing the dysregulation in calcium levels in the central nervous system by administering compounds such as MEM 1003 may have the potential for altering the cyclical course or progression of bipolar disorder.

MEM 1003 is the (+)-enantiomer of a dihydropyridine that has been optimized for central nervous system activity. It inhibits L-type Ca2+ channels and within the anticipated human dosing range has more benign cardiovascular effects than other DHP L-Type calcium channel modulators.

ELIGIBILITY:
Inclusion Criteria:

* bipolar I disorder with acute manic or mixed episode, with or without psychotic features
* YMRS score of at least 20
* history of at least one previous manic or mixed episode requiring treatment in the last 10 years

Exclusion Criteria:

* history of failing to respond to treatment with two or more adequate trials of approved anti-manic medications for the current episode
* Axis I or Axis II disorder (other than bipolar I disorder) that requires treatment or has been the primary subject of treatment in the past 3 months
* defined substance abuse or dependency within the 3 months
* schizophrenia, schizoaffective disorder, delusional disorder, mental retardation or pervasive developmental disorder
* suicidal or danger to others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-09; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Response rate at Day 21

SECONDARY OUTCOMES:
Change from baseline to Day 21 in other efficacy measures and safety

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Murray, MD, PhD, Study Director — Memory Pharmaceuticals Corp
Locations (18):
- United States (18):
  - Little Rock, Arkansas
  - Garden Grove, California
  - Riverside, California
  - San Diego, California
  - Torrance, California
  - Bradenton, Florida
  - Fort Lauderdale, Florida
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Willingboro, New Jersey
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Bellaire, Texas
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - Kirkland, Washington